CLINICAL TRIAL: NCT02168517
Title: Obesity, Pain and Fertility: is There Any Association?
Brief Title: Correlation of Pain, Obesity and Fertility Potential.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Sponsor
Other Study IDs: N-20140025
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Overweight and Obesity
Keywords: Obesity; Pain; Fertility
MeSH Terms: conditions — Overweight; Obesity; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — A research biobank will be established during the project period. Majority of each sperm sample will be analyzed immediately but approximately 250 ul seminal plasma will be frozen and later analyzed at Aalborg University Biotechnology Department.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Group I: Overweight osteoarthritis patients
- Group II: Normal weight osteoarthritis patients.
- Group III: Overweight healthy men.
- Group IV: Normal weight healthy men.

SUMMARY:
The overall aim of the study is to investigate if patients with musculoskeletal chronic pain have reduced semen quality in comparison with age matched healthy controls. Secondly, the aim is to investigate whether overweight with or without chronic pain are related to reduced semen quality. We will investigate semen quality in obese chronic pain patients, normal weight chronic pain patients and in obese and normal weight healthy controls.

DETAILED DESCRIPTION:
Obesity is associated with several disorders including chronic musculoskeletal pain. For example obesity has been implicated in the development or progression of low back pain and knee osteoarthritis. The mechanism by which obesity causes lumbar back pain is poorly understood, but the contribution of both mechanical and system factors is likely. Direct mechanical stress on the intervertebral discs and adjacent structures are suspected to be mechanisms through which obesity affects the spine, leading to subsequent low back pain. The link between obesity and knee osteoarthritis has also been demonstrated, but potential factors underlying the association of obesity with knee osteoarthritis has not entirely been elucidated.

It is a well-known fact that obesity leads to an excess load on the joint, increased cartilage turnover, increased collagen type 2 degradation products and increased risk of degenerative meniscal lesions. Although all of these factors have been proposed to lead to knee osteoarthritis, no causal relationship has been demonstrated.

ELIGIBILITY:
Inclusion Criteria:

* Men between 18-45 years with low back pain or knee pain recruited among referees to the orthopaedic outpatient clinics at Aalborg University Hospital
* Pain more than 3 months
* Patients can be on a daily use of Paracetamol 1 gram x 4, NSAID x 3-4 or combined
* Patients will be included regardless of their BMI but will be put in their respective BMI subgroup after the required measurements have been taken
* Regarding low back pain the LBPRS >9, knee pain the KOOS <75 (0-100, i.c. 100 = no problems)
* Healthy men in the age 18-45 years (matched with enrolled patients)

Exclusion Criteria:

* Malignancy
* Ongoing infection
* Drug addiction defined as the use of cannabis, opioids or other psycho drugs
* Previous neurologic, musculoskeletal or mental diseases
* Lack of ability to cooperate
* Pain rating
* Patients with a pain rate below 3
* Medication
* Patients taking Morphine drugs

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Progressive motility | 6 months
  Progressive motility as in the world health organization lower reference limits for sperm quality.

SECONDARY OUTCOMES:
Pain | 6 months
  The patients will be tested for their pain in terms of intensity and quality. Intensity will be rated on a visual analogue scale (VAS 0-10) for ongoing pain. Pressure pain will be measured by application of a handheld pressure algometer. A validated Danish version of short form McGill Pain Questionnaire will be given to evaluate the quality of pain. In addition, distribution of pain will be mapped by drawing on a body chart.

CONTACTS AND LOCATIONS:
Overall Officials: Sten Rasmussen, M.D., Study Director — Clinic for Neuro- and Orthopaedic Diseases, Aalborg University Hospital; Hans I. Nielsen, PhD, Study Director — Department of Health Science and Technology, Aalborg University; Fereshteh Dardmeh, PhD stud., Principal Investigator — Department of Health Science and Technology, Aalborg University; Parisa Gazerani, PhD, Study Chair — Department of Health Science and Technology, Aalborg University; Hiva Alipour, PhD stud., Study Chair — Department of Health Science and Technology, Aalborg University
Locations (1):
- Clinic for Neuro- and Orthopaedic Diseases, Aalborg University Hospital, Aalborg, Denmark